CLINICAL TRIAL: NCT03301571
Title: Response in Right Ventricular Function to Change in Afterload, Preload and Inspired Oxygen in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Right Ventricular Echocardiography in caRdiac SurgEry
Acronym: ReVERSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lars Grønlykke, Principal investigator, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17005565
Record Dates: First submitted 2017-09-19; First posted 2017-10-04 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Right Ventricular Dysfunction
Keywords: Coronary artery bypass graft; Echocardiography
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Intervention Model Description: All patients will receive the same interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): All patients will receive the treatment (CABG) and postoperatively three different interventions:
  1. Change in preload and afterload
  2. Change in inspired oxygen
  3. Change in pacemaker modes
  Interventions: Other: Change in preload and afterload; Other: Inspired oxygen; Other: Pacemaker mode

INTERVENTIONS:
Other: Change in preload and afterload — Afterload: Three levels of positive end-expiratory pressure (PEEP) will be examined post-operatively: 0 cm H20, 5 cm H2O, 10 cm H2O Preload: Trendelenburg position for 5 minutes will be investigated
Other: Inspired oxygen — Following fractions of inspired O2 will be investigated: 0.5 and 1.0 for 10 minutes respectively
Other: Pacemaker mode — Following pacemaker settings will be investigated: Atrioventricular pacing 10 bpm over the patients' intrinsic rhythm, atrial pacing 10 bpm over the patients' intrinsic rhythm, ventricular pacing 10 bpm over the patients' intrinsic rhythm

SUMMARY:
Postoperative right ventricular (RV) dysfunction increases mortality and risk of cardiac failure after cardiac surgery substantially. A comprehensive understanding of this condition is paramount in order to achieve success in treatment and early diagnosis.

This study has two main aims.

Perioperative aim:

To investigate correlations between changes in echocardiographic measurements and hemodynamic changes at baseline and following coronary artery bypass graft (CABG) surgery.

Postoperative aim:

To evaluate changes in haemodynamics and echocardiographic parameters during separate physiological interventions (increase in preload/afterload, oxygen fraction, pacing modes (AAI/DDD/VVI)).

DETAILED DESCRIPTION:
Clinical procedure:

For the operation standard procedures for anaesthesia, surgery and cardiopulmonary bypass will be used. This includes installment of a pulmonary artery catheter and performing a transesophageal echocardiography. For the purpose of this study additional TEE images and a transthoracic echocardiography (TTE) will be obtained in order to correlate different echocardiographic indices with haemodynamic measurements and investigate any differences between TTE and TEE measurements.

Transthoracic echocardiography (TTE):

Basic TTE will be performed after anaesthesia induction, before surgery commences and repeated immediately after arrival at the ICU.

Image acquisitions from TTE:

* 2D apical 4-chamber view for right ventricular fractional area change (RVFAC)
* M-mode tricuspid annular plane systolic excursion (TAPSE).
* M-mode lateral mitral annular plane systolic excursion (MAPSE) measurements

Transoesophageal echocardiography (TEE):

After probe placement and before commencing surgery a TEE will be performed. The probe will be left in place during surgery for continuous imaging. Standard views used for patient treatment will be acquired in accordance with the requirements of the treating anaesthesiologist and surgeon.

Additional views will be added in order to obtain standard 2D measures, M-mode measures, spectral doppler measures, myocardial doppler tissue imaging, strain and 3D measures of RV function.

Measurements will be performed at different stages throughout surgery following a period of relative hemodynamic stability defined as: 1 minute of no more than 10 beats/min variation in heart rate, maximum variation of 10 mmHg in mean arterial pressure, maximum variation of 3 mmHg in central venous pressure and no change in administration of vasoactive drugs. If hemodynamic stability cannot be achieved an annotation comment will be entered.

Time points for echocardiography:

TEE will be performed at four different time points during and immediately after surgery:

Stage 1: After induction of anaesthesia. Stage 2: After full sternotomy Stage 3: After completion of cardiopulmonary bypass Stage 4: Immediately after arrival at the ICU and will be repeated after each intervention

Interventions Each intervention will be investigated separately and before each intervention the patient will return to hemodynamic baseline.

Trendelenburg position for 5 minutes will be investigated. Following positive end-expiratory pressures will be investigated: 0 cm H2O, 5 cm H2O and 10 cm H2O.

Following fractions of inspired O2 will be investigated: 0.5 and 1.0 for 10 minutes at each setting.

Following pacemaker settings will be investigated: Atrioventricular pacing 10 bpm over the patients' intrinsic rhythm, atrial pacing 10 bpm over the patients' intrinsic rhythm, ventricular pacing 10 bpm over the patients' intrinsic rhythm

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass graft patients
* Normal left ventricular function defined as LVEF over 50 % on TTE preoperatively

Exclusion Criteria:

* Pre-existing right ventricular malformations
* Severe right ventricular impairment preoperatively
* Pre-existing non-sinus rhythm
* Pre-existing mitral valve stenosis or severe regurgitation
* Pre-existing pulmonary hypertension
* Pre-existing tricuspid valve stenosis or severe regurgitation
* Patients with contraindication to TEE probe placement such as oesophageal stricture or obstruction
* Patients with contraindication to Swan-Ganz catheter placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Change in right ventricular function during CABG assessed with TAPSE | During a standard CABG operation
  Assessing the change in RV function during CABG surgery

SECONDARY OUTCOMES:
Right ventricular function assessed with TAPSE after each intervention | Immediate postoperative period
  Change in TAPSE after each intervention
Change in cardiac output measured with Swan-Ganz during CABG | During a standard CABG operation
  Cardiac output measured with the thermodilution technique
Change in cardiac output measured with Swan-Ganz after each intervention | Immediate postoperative period
  Cardiac output measured with the thermodilution technique
Response in right ventricular function parameter S' to each intervention | Immediate postoperative period
  Change in S'
Response in right ventricular function parameter S' during CABG | During a standard CABG operation
  Change in S'
Response in right ventricular function parameter Tei index to each intervention | Immediate postoperative period
  Change in Tei index
Response in right ventricular function parameter Tei index during a standard CABG operation | During a standard CABG operation
  Change in Tei index
Response in right ventricular function parameter RVFAC to each intervention | Immediate postoperative period
  Change in RVFAC
Response in right ventricular function parameter RVFAC during a standard CABG operation | During a standard CABG operation
  Change in RVFAC
Response in left ventricular function parameter MAPSE to each intervention | Immediate postoperative period
  Change in MAPSE
Response in left ventricular function parameter MAPSE during a standard CABG operation | During a standard CABG operation
  Change in MAPSE
Response in right ventricular function parameter strain % to each intervention | Immediate postoperative period
  Change in strain %
Response in right ventricular function parameter strain % during a standard CABG operation | During a standard CABG operation
  Change in strain %
Response in right ventricular function parameter strain rate to each intervention | Immediate postoperative period
  Change in strain rate
Response in right ventricular function parameter strain rate during a standard CABG operation | During a standard CABG operation
  Change in strain rate
Response in right ventricular function parameter RV size to each intervention | Immediate postoperative period
  Change in RV size
Response in right ventricular function parameter RV size during a standard CABG operation | During a standard CABG operation
  Change in RV size
Response in right ventricular function parameter pulmonary artery flow velocity to each intervention | Immediate postoperative period
  Change in flow velocity in pulmonary artery
Response in right ventricular function parameter pulmonary artery flow velocity during a standard CABG operation | During a standard CABG operation
  Change in flow velocity in pulmonary artery
Response in right ventricular function parameter RVEF to each intervention | Immediate postoperative period
  Change in RVEF measured with 3D echo
Response in right ventricular function parameter RVEF during a standard CABG operation | During a standard CABG operation
  Change in RVEF measured with 3D echo
Response in right ventricular function parameter RVEF during CABG | Immediate postoperative period
  Change in RVEF measured with 3D echo
Change in cardiac output measured with Swan Ganz in response during a standard CABG operation | During a standard CABG operation
  Following each intervention in the postoperative period cardiac output will be measured with the thermodilution technique.
Change in cardiac output measured with Swan Ganz in response to each intervention | Immediate postoperative period
  Following each intervention in the postoperative period cardiac output will be measured with the thermodilution technique.
Change in hemodynamic pressures in response to each intervention | Immediate postoperative period
  Following each intervention in the postoperative period hemodynamic pressures will be measured with the Swan Ganz catheter
Change in hemodynamic pressures during a standard CABG operation | During a standard CABG operation
  Following each intervention in the postoperative period hemodynamic pressures will be measured with the Swan Ganz catheter

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grønlykke, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No